CLINICAL TRIAL: NCT06236841
Title: A Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Food Effects of XH-S004 Single and Multiple Ascending Doses in Healthy Volunteers
Brief Title: A Phase I Study of XH-S004 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: S-INFINITY Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-S004-101
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XH-S004 (Experimental): Participants will receive XH-S004 as per assigned treatment regimen on scheduled days. Starting dose in single asceding dose: 5 mg.
  Interventions: Drug: XH-S004 tablet
- XH-S004 placebo tablet (Placebo Comparator): Participants will receive matching placebo as per assigned treatment regimen on scheduled days.
  Interventions: Drug: XH-S004 placebo tablet

INTERVENTIONS:
Drug: XH-S004 tablet — XH-S004 tablets will be administered orally as per assigned treatment regimen on schedualed days.
  Arms: XH-S004
Drug: XH-S004 placebo tablet — XH-S004 placebo tablet (matched) will be administered orally as per assigned treatment regimen on schedualed days.
  Arms: XH-S004 placebo tablet

SUMMARY:
This is a phase I, randomised, double-blind placebo-controlled, 3-part study to assess the safety, tolerability, pharmacokinetics and food effect of single and multiple oral doses of XH-S004 in healthy volunteers.

ELIGIBILITY:
Inclusive criteria:

1. Healthy male and female subjects, 18 to 45 years of age (inclusive) at Screening.
2. Male body weight no less than 50 kilogram (Kg), Female body weight no less than 45 Kg, and body mass index (BMI) between 16.0 and 26.0 kg/m2 (both inclusive).
3. Medically healthy without no clinically significant abnormalities on the basis of inquiry, vital signs, physical examination, 12-lead electrocardiogram (ECG), laboratory tests (hematology, serum chemistry, coagulation function and urinalysis, etc,) , and chest X-ray, etc,.
4. Participants must be able to understand the procedures and methods of this study, and voluntarily take part in this study, and communicate well with investigators, and comply with requirements throughout the study, and sign the informed consent form (ICF).
5. Subjects must guarantee and agree to take effective contraceptive methods (example, condom and intrauterine device) other than oral medication from 14 days prior to signing ICF to 30 days after last dose, and have no plan to donate sperm and ovum during the study.

Exclusive criteria:

1. Pregnant or lactating woman, or woman with a positive pregnancy test.
2. Participants who are suspected or confirmed to be allergic to any ingredients of investigational product, or participants who are allergic, or have a drug allergy history or specific allergic disorders (asthma, urticaria, eczema, etc.).
3. Participants with a medical history or a presence of significant cardiovascular, pulmonary, endocrine, urinary/reproductive, gastrointestinal, dermatologic, immunologic, hematological, neurological, psychiatric and infectious diseases or abnormalities; Or any acute, chronic disease or physiological condition that could interfere with the study results.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-26 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
To access the incidence and severity of adverse events (AEs), serious AEs and abnormalities on laboratory tests [Safety and Tolerability] of single ascending oral dose of XH-S004 in healthy adults. | Approximately 1~2 weeks.
  The incidence and severity of adverse events (AEs) , serious AEs and abnormalities on laboratory tests.
To access the incidence and severity of adverse events (AEs), serious AEs and abnormalities on laboratory tests [Safety and Tolerability] of multiple ascending oral dose of XH-S004 in healthy adults. | Approximately 2 months.
  The incidence and severity of adverse events (AEs) , serious AEs and abnormalities on laboratory tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing LuHe Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No